CLINICAL TRIAL: NCT04292860
Title: Reverse Axillary Mapping as a Lymphedema Prevention Strategy in Breast Radiation Treatment Planning
Brief Title: Reverse Axillary Mapping in Breast Radiation Treatment Planning
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator decided not to move forward with the study
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1934
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer; Lymphedema
Keywords: Lymphedema; Axillary Reverse Mapping; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Pts: Post-operative (lumpectomy or mastectomy) female breast cancer patients who will receive radiation to the whole breast or chest wall and the regional nodes.

SUMMARY:
The goal of this prospective study is to investigate the role of axillary reverse mapping (ARM) in radiation therapy planning of patients with breast cancer. Lymphedema is a common side effect after surgery and radiation therapy for breast cancer. The use of ARM is becoming more routine in surgery to differentiate the upper extremity lymphatics (UELs) from the breast axillary drainage to preferentially spare the UELs and reduce the rates of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* De novo presentation of post-operative (lumpectomy or mastectomy) female breast cancer patients to receive radiation to the whole breast or chest wall and the regional nodes. Patients who have received a sentinel lymph node (SLN) biopsy or an axillary lymph node dissection (ALND) will be eligible.
* Greater than or equal to 18 years of age (no upper age limit).
* Informed consent obtained.

Exclusion Criteria:

* Prisoners.
* Patients with metastatic breast cancer.
* Documented allergy to iodinated contrast
* Prior breast or axillary surgeries or radiation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-operative (lumpectomy or mastectomy) female breast cancer patients who will receive radiation to the whole breast or chest wall and the regional nodes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Delineation of the upper extremity lymphatics (UEL) during the radiation treatment planning process using axillary reverse mapping (ARM) | Baseline to 1 year
  ARM uses dye to track lymphatic flow of the upper extremities.We hypothesize that iodinated contrast injected into the upper inner arm (same site that surgeons inject during ARM) 15 minutes before the time of CT simulation will similarly be able to track the UELs. We will contour the visible iodinated dye and will measure if that anatomically correlates with the general known location of the UELs. Two radiation oncologists will independently determine if they can delineate the UELs. If both radiation oncologists can identify and contour the UELs in a reproducible fashion, we will code the patient as "UEL identified." If one or both physicians are either not able to identify the UEL on CT images or the contoured UEL structures are significantly different from each other, we will code the patient as "UEL not identified."

SECONDARY OUTCOMES:
Dosimetric endpoint | Baseline to 1 year
  We will measure the Dmax, Dmin, Dmean, D25%, and D75%. Dmax is the maximum dose (in units of Gray) delivered to the UEL, while Dmin is the minimum dose and Dmean is the mean dose. D25% and D75% are the minimum dose delivered to 25% and 75% of the UEL, respectively. We will also look at the percent of theoretical radiation plans that could be safely modified. This will be a binary outcome: either the plan can be modified safely, or it cannot.
Lymphedema rate | Baseline to 5 years post-treatment
  We will measure the lymphedema rates before the start of radiation and at 6 months, 12 months, 24 months, 36 months, and 60 months after the end of radiation therapy. Arm circumference will be measured 15 cm above the medial epicondyle (upper arms) and 15 cm below the medial epicondyle (lower arms. An increase in arm circumference of at least 10% in the lower arm or the upper arm, or both, compared with the contralateral arm at the same time-point will be considered clinically significant lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Casey, Principal Investigator — UNC Chapel Hill